CLINICAL TRIAL: NCT04818593
Title: A Sibling Oocyte Study- Comparison of ZyMotTM Microfluidics Device to Density Gradient for Sperm Selection During ICSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-00021
Record Dates: First submitted 2021-03-25; First posted 2021-03-26 (Actual); Results first posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: ART
Keywords: ICSI
MeSH Terms: interventions — Centrifugation, Density Gradient

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- ZyMot Separation (Experimental): Treatment
  Interventions: Device: ZyMot Multi Sperm Separation Device (850 ul)
- Density Gradient Centrifugation (Active Comparator): Control
  Interventions: Other: Density Gradient Centrifugation

INTERVENTIONS:
Device: ZyMot Multi Sperm Separation Device (850 ul) — 850 uL of untreated semen will be directly deposited into the inlet port of the ZyMotTM Multi device, followed by placement of 750 uL culture medium in the outlet port and throughout the upper collection chamber. The device will then be incubated in a humidified 37C CO2 incubator for 30 minutes. During incubation, the healthiest and most motile sperm will swim through the microporous filter and into the upper collection chamber, where they will be recovered via the outlet port. 500 uL of the sperm sample will be removed and placed in a separate tube for analysis and insemination.
  Arms: ZyMot Separation
Other: Density Gradient Centrifugation — Density gradient centrifugation will be performed using a one-layer preparation of 90% Isolate in 15 mL conical tubes. Semen will be layered over 1 mL of gradient and then centrifuged for 15 min at 300xg. The supernatant will be removed and discarded. The sperm pellet will be washed by mixing with Multipurpose Handling Medium Complete and centrifuging the sample for 5 min at 400xg. After the wash, the supernatant is removed and discarded and the pellet is re-suspended in culture medium, assessed for sperm parameters, and held at room temperature until insemination.
  Arms: Density Gradient Centrifugation

SUMMARY:
The primary objective of this study is to evaluate whether the percentage of good quality embryo formation following Intracytoplasmic Sperm Injection (ICSI) is improved with the use of ZyMot method of microfluidic sperm separation compared to density gradient.

DETAILED DESCRIPTION:
During an in vitro fertilization (IVF) cycle, eggs are removed from a woman's ovaries via a minor surgical procedure and are inseminated with sperm in order to create embryos. The insemination process can be via standard IVF or intracytoplasmic sperm injection (ICSI.) Standard IVF is the process of placing thousands of sperm in a culture dish with one or more eggs and allowing them to interact on their own. ICSI is the process by which one sperm is directly injected into each egg.

Prior to using the sperm for insemination, a semen sample is processed and washed in order to obtain the healthiest sperm. A standard sperm preparation procedure is density gradient, in which the sperm is spun via centrifugation and separated from the seminal fluid. An alternate method is via microfluidics, by which the sperm swim up a microfluidic gradient created by a microporous filter between two chambers of a device. Sperm that are capable of navigating through this filter and reaching the end chamber are presumed to be the healthiest sperm. There is some data revealing that ZyMot microfluidics yields healthier sperm compared to the density gradient technique.

The aim of the study is to evaluate whether good quality embryo formation is any different following insemination with sperm separated by microfluidics compared to density gradient.

On the day of oocyte retrieval, the sperm sample will be split between the two different processing methods: density gradient and ZyMot microfluidics. In the event that there are 6 or more mature oocytes and ICSI will be used for insemination, half of the oocytes will be inseminated with sperm processed by density gradient and half with sperm processed by ZyMot microfluidics. The percentage of good quality embryo formation will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria for Patients:

1. Patient(s) over 18 years of age
2. Patient(s) capable of providing informed consent
3. Use or possible use of ICSI for oocyte insemination
4. At least 6 mature oocytes at time of insemination via ICSI

Exclusion Criteria for Patients:

1. Patient under 18 y/o
2. Patients not capable of providing informed consent
3. Use of IVF for insemination
4. Less than 6 mature oocytes at time of rertrieval
5. Anonymous donor sperm source
6. Surgically retrieved sperm
7. Sperm sample not sufficient for use with ZyMot device

Inclusion Criteria for Donors:

1. Donor(s) over 18 years of age
2. Donor(s) capable of providing informed consent
3. Use of ejaculate sperm, fresh or frozen, for insemination
4. Sufficient sperm for use of ZyMot

Exclusion Criteria for Donors:

1. Anonymous donors

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2021-06-18 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2021-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rani Fritz, DO, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Reproductive Specialists of NY, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared at the discretion of the PI.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data at the discretion of the PI. Requests should be directed to Rani.Fritz@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The trial enrolled 108 unique individuals grouped into 54 patient/sperm-source dyads. Each enrolled dyad produced oocyte units. Oocytes from the same dyad were assigned to the density gradient (control) arm, ZyMot (treatment) arm, or both depending on the criteria met by the oocyte units, meaning the same 54 dyads were assigned to both study arms. Dyads who produced insufficient samples for ZyMot processing were withdrawn.
Units Other Than Participants: Oocytes
Groups:
- ZyMot Separation Device (Treatment): 850 uL of untreated semen will be directly deposited into the inlet port of the ZyMotTM Multi device, followed by placement of 750 uL culture medium in the outlet port and throughout the upper collection chamber. The device will then be incubated in a humidified 37C CO2 incubator for 30 minutes. During incubation, the healthiest and most motile sperm will swim through the microporous filter and into the upper collection chamber, where they will be recovered via the outlet port. 500 uL of the sperm sample will be removed and placed in a separate tube for analysis and insemination.
  Control: Density Gradient Centrifugation: Density gradient centrifugation will be performed using a one-layer preparation of 90% Isolate in 15 mL conical tubes. Semen will be layered over 1 mL of gradient and then centrifuged for 15 min at 300xg. The supernatant will be removed and discarded. The sperm pellet will be washed by mixing with Multipurpose Handling Medium Complete and centrifuging the sample for 5 min at 400xg. After the wash, the supernatant is removed and discarded and the pellet is re-suspended in culture medium, assessed for sperm parameters, and held at room temperature until insemination.
- Density Gradient Centrifugation (Control): Density gradient centrifugation will be performed using a one-layer preparation of 90% Isolate in 15 mL conical tubes. Semen will be layered over 1 mL of gradient and then centrifuged for 15 min at 300xg. The supernatant will be removed and discarded. The sperm pellet will be washed by mixing with Multipurpose Handling Medium Complete and centrifuging the sample for 5 min at 400xg. After the wash, the supernatant is removed and discarded and the pellet is re-suspended in culture medium, assessed for sperm parameters, and held at room temperature until insemination.
Period: Overall Study
Arm/Group | ZyMot Separation Device (Treatment) | Density Gradient Centrifugation (Control)
Started | 54; 231 Oocytes | 54; 225 Oocytes
Completed (Oocyte units were assigned to density gradient and/or ZyMot microfluidics insemination techniques depending on how they met study criteria. Sperm samples that were insufficient for ZyMot processing were not processed and the corresponding participant dyad was withdrawn from the study. The number of oocyte units that started the study for each arm is equal to the number completed, as the unit number (oocytes) is not known for the cycles that were withdrawn from the study and cannot be calculated.) | 34; 231 Oocytes | 34; 225 Oocytes
Not Completed | 20; 0 Oocytes | 20; 0 Oocytes
Not completed — Low Oocyte Yield | 8 | 8
Not completed — Not ICSI Insemination | 7 | 7
Not completed — Poor Sperm Quality | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Conversion to IUI due to low response | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline data were collected only on the level of the participants (not oocyte units). The overall number of baseline participants represents individuals (n = 66) from dyads that completed the trial. Information from one dyad (2 individuals) were not collected.
Groups:
- Study Population: Individuals in patient/sperm-source dyads with oocyte units that were analyzed.
Arm/Group | Study Population
Number analyzed (Participants) | 66
Age, Continuous [Median (Standard Deviation); unit: years] | 36.9 (0.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 65

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Good Quality Blastocyst Formation
Description: Good quality embryos will be defined as blastocyst stage embryos on day 5 or 6 of culture with an overall quality grade of good or fair. Embryo morphology assessment includes two parts: an Overall Grade and the Stage. Grading is a subjective assessment of the overall quality of the embryo as good, fair, or poor, and is based on assessment of certain characteristics of the embryo, such as fragmentation, symmetry, inner cell mass (ICM) quality and trophectoderm quality. The percentage will be reported for both arms (ZyMot compared to density gradient).
Time Frame: Culture Day 5 or 6
Population: Participants refer to dyads. Information form one of the completed dyads was not collected.
Measure: Mean (Standard Deviation); unit: percentage of embryos
Units Other Than Participants: Oocytes
Arm/Group | ZyMot Separation | Density Gradient Centrifugation
Number analyzed (Participants) | 33 | 33
Number analyzed (Oocytes) | 231 | 225
percentage of embryos | 51.4 (5.1) | 51.7 (5.4)

ADVERSE EVENTS:
Time Frame: Up to 2 weeks post-embryo transfer
Description: PI monitored for adverse events/serious adverse events/all-cause mortality. The number of participants at Risk (n = 33) represents the number of dyads assigned to each intervention for whom adverse event/serious adverse event/all-cause mortality data were collected.
Arm/Group | ZyMot Separation | Density Gradient Centrifugation
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 0/33 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-17): https://cdn.clinicaltrials.gov/large-docs/93/NCT04818593/Prot_SAP_000.pdf